CLINICAL TRIAL: NCT04631952
Title: A Randomised Controlled Trial of Online Exercise Intervention for Psychosis Patients Receiving Residential Care in Hong Kong
Brief Title: Online Exercise Intervention for Psychosis Patients Receiving Residential Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Yi-Nam Suen, Research Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SMI_exercise_RCT
Record Dates: First submitted 2020-11-16; First posted 2020-11-17 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Psychosis
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online exercise (Experimental): SMS messages on encouraging active lifestyle plus an online exercise video
  Interventions: Behavioral: Online exercise
- SMS message (Active Comparator): SMS messages on encouraging active lifestyle
  Interventions: Behavioral: SMS message

INTERVENTIONS:
Behavioral: Online exercise — SMS messeages on encouraging active lifestyle and online exercise video will be sent to the participant weekly for 8 weeks.
  Arms: Online exercise
Behavioral: SMS message — SMS messeages on encouraging active lifestyle will be sent to the participant weekly for 8 weeks.
  Arms: SMS message

SUMMARY:
The main objective of this randomised controlled trial (RCT) is to investigate the immediate and long-term effectiveness of 8-week online exercise intervention for people with psychosis receiving residential care.

DETAILED DESCRIPTION:
The effect will also be evaluated after 6-month and 12-month, anticipate seeing the maintenance of physical activity throughout a year of time.

The secondary objective of this RCT is to investigate if the exercise intervention will be effective in improving the clinical symptoms, cognitive functioning and social functioning of the subjects, and to see if the improvement can be maintained (or improve) over a longer period of time (i.e., 6-month and 12-month).

ELIGIBILITY:
Inclusion Criteria:

* Based on the Fifth version of the Diagnostic and Statistical Manual of Mental Disorders diagnosis to have schizophrenia and related psychotic disorders
* Have the ability to understand Chinese
* Able to give informed consent

Exclusion Criteria:

* Severe physical illness (Myocardial Infarction, Hypertension, Fracture, Spinal problems in which exercise may be contraindicated), and seizure disorders.
* Comorbid substance dependence
* Unstable psychotic symptoms
* Any history of brain trauma or organic brain disease
* Known history of intellectual disability or special school attendance
* Other mental conditions that requires other treatment priorities, e.g., suicidal risk.
* Other medical conditions that severely limits participation, comprehension, or adherence to the treatment or assessment e.g., epilepsy, dementia, terminal medical illness.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Exercise level | 6 months and 12 months
  Measured by the International Physical Activity Questionnaire, a higher MET calculated from the scale indicates a higher exercise level

SECONDARY OUTCOMES:
Severity of psychotic symptoms | 6 and 12 months
  Measured by the Positive and Negative Syndrome Scale, a higher score indicates a more severe level of psychotic symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Yi Nam Suen, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No